CLINICAL TRIAL: NCT03013816
Title: Increasing Donor Designation Rates in Teenagers: Effectiveness of a Driver's Education Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, James Rodrigue, Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015P000063
Record Dates: First submitted 2016-12-29; First posted 2017-01-09 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Organ Donor Registration; Organ Donation Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Testimonial Messaging (Experimental): This video features four personal testimonials with strong emotional appeal, including an adolescent kidney transplant recipient, a pediatric liver transplant recipient, a young adult kidney transplant candidate, and an adolescent whose twin brother was a deceased organ donor. There are minimal facts about transplantation or donation.
  Interventions: Behavioral: Organ Donation Education: Testimonial Messaging
- Informational Messaging (Experimental): This video mirrors common educational campaigns and included segments of HRSA's animated video, Organ Donation and Transplantation: How Does it Work? The IM video presents facts about donation, including the current supply-demand problem in transplantation, common reasons for/against donor designation, donation myths, and the importance of communicating with parents about donation. Information about how to register as a donor is also included. The video contains no personal testimonials.
  Interventions: Behavioral: Organ Donation Education: Informational Messaging
- Blended Messaging (Experimental): This video features four personal testimonials with strong emotional appeal, including an adolescent kidney transplant recipient, a pediatric liver transplant recipient, a young adult kidney transplant candidate, and an adolescent whose twin brother was a deceased organ donor. There are minimal facts about transplantation or donation.
  Interventions: Behavioral: Organ Donation Education: Blended Messaging

INTERVENTIONS:
Behavioral: Organ Donation Education: Testimonial Messaging — The testimonial messaging video intervention will be shown
  Arms: Testimonial Messaging
Behavioral: Organ Donation Education: Informational Messaging — The informational messaging video intervention will be shown
  Arms: Informational Messaging
Behavioral: Organ Donation Education: Blended Messaging — The blended messaging video intervention will be shown
  Arms: Blended Messaging

SUMMARY:
Four aims were pursued: (1) Evaluate the effectiveness of video messaging on adolescent donor designations in comparison to a regionally-matched historical comparison group of adolescents; (2) Compare the differential effectiveness of three commonly-used donation messaging strategies (informational, testimonial, and blended) on donor designations; (3) Examine the impact of donation messaging on changes in secondary outcomes (donation engagement, knowledge, attitudes, beliefs, likelihood of donor designation, discussion with a parent) before and after video intervention; and (4) Assess the commitment of parents to follow their adolescent's donation wishes in the event of death. Our central hypotheses were that integrating donation video messaging into driver education classes would generate a higher proportion of donor designations compared to a historical comparison group and that blended video messaging (informational + testimonials) would yield a higher proportion of donor designations and more change in secondary outcomes.

ELIGIBILITY:
Criteria for Classrooms:

Classroom eligibility criteria included: (a) driver education conducted in English, and (b) instructor agreement not to provide or discuss donation information beyond the study video.

Criteria for Adolescent Participants:

Inclusion Criteria:

* Enrolled in driving school class
* English speaking
* Adolescent assent
* Parental permission to participate

Exclusion Criteria:

* Prior participation in a driver's education class in which organ donation education was provided
* Parent permission form not signed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Organ Donation Registration | 6 months
  The primary outcome was donor designation (yes-no) at time of obtaining first driver's license post-intervention. We provided the name, date of birth, last four digits of social security number, residential address, and study identification number of each adolescent to the Massachusetts DoT, which then returned to us a data file containing the donor designation status for each study identification number. For the regionally-matched historical comparison group, the DoT provided a de-identified data file of all adolescents who obtained their first driver's license in the six months prior to study enrollment at six motor vehicle offices.

SECONDARY OUTCOMES:
Organ Donation Knowledge and Attitudes | 1 week
  Immediately before, shortly after, and 1 week following video messaging exposure, adolescents completed a questionnaire to assess the following donation constructs: engagement (2 questions -- 1-10 scale), knowledge (3 questions -- correct/incorrect total score range 0-3), general attitude (1 question), beliefs (4 questions -- strong disagree-strongly agree scale), designation likelihood (1 question -- 1-10 scale), and willingness to communicate donation decision to a parent (1 question -- 1-10 scale). Adolescents received a $5 gift card for each survey completed.
Parental Commitment | 6 months
  One week following the adolescent's exposure to the donation video, we mailed parents a brief questionnaire that included questions about their donor designation status (Yes/No), general donation attitude (1 question -- 1-10 scale), any communication with their adolescent about his/her donor designation intention (Yes/No), and likelihood of following their adolescent's wishes about donation (1 question -- 1-10 scale).

CONTACTS AND LOCATIONS:
Overall Officials: James Rodrigue, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigue JR, Boger M, DuBay D, Fleishman A. Increasing Organ Donor Designation Rates in Adolescents: A Cluster Randomized Trial. Am J Public Health. 2019 Sep;109(9):1273-1279. doi: 10.2105/AJPH.2019.305178. Epub 2019 Jul 18. PMID 31318603